CLINICAL TRIAL: NCT04444206
Title: Prevention of Preterm Birth by Universal Screening With Ultrasound Measurement of the Consistency Index and Length of the Uterine Cervix in Women With a Single
Brief Title: Prevention of Preterm Birth by Screening of the Consistency Index and Length of the Uterine Cervix in Women With a Single Pregnancy
Acronym: PreBirthCerv
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Prof. Pasquale De Franciscis, Associate Professor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 8451
Record Dates: First submitted 2020-06-20; First posted 2020-06-23 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Pregnancy, High Risk; Preterm Birth; Cervix; Pregnancy; Obstetric Labor, Premature; Obstetric Labor Complications; Pregnancy Complications
Keywords: ultrasound
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature; Obstetric Labor Complications; Pregnancy Complications

STUDY DESIGN:
Intervention Model Description: This is a prospective, non-pharmacological, non-profit interventional study on women with single pregnancy without a history of previous preterm spontaneous birth. Cervical lenght (CL) and Consistence Cervical Index (CCI) will be assessed by transvaginal ultrasound. CL and CCI measurements will be performed in the first trimester, between 11 and 13 weeks + 6 days, in the second trimester, between 19 and 22 weeks and in the third trimester between 29 and 32 weeks during routine ultrasound examinations for monitoring of pregnancy, in accordance with current national guidelines.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CL and CCI screening (Experimental): The Cervical lenght (CL) and the Consistence Cervix Index (CCI) will be evaluated by transvaginal ultrasound. CL and CCI measurements will be expected in the first trimester, between 11 and 13 weeks + 6 days, in the second trimester, between 19 and 22 weeks and in the third trimester between 29 and 32 weeks during the ultrasound examinations required by the monitoring routine of pregnancy, in accordance with current national guidelines.
  Interventions: Procedure: Transvaginal ultrasound cervical length screening
- No CL and CCI screening (No Intervention): The investigators collect data of these pregnant women without any additional ultrasound examination

INTERVENTIONS:
Procedure: Transvaginal ultrasound cervical length screening — Cervical lenght and Consistence Cervical Index measurements performed, between 11 and 13 weeks + 6 days, in the , between 19 and 22 weeks and i between 29 and 32 weeks during the ultrasound examinations required by the monitoring routine of pregnancy.
  Arms: CL and CCI screening

SUMMARY:
Preterm birth (PTB) is the major cause of perinatal morbidity and mortality. Worldwide, about 15 million babies are born too soon every year, causing 1.1 million deaths, as well as short- and long-term disability in countless survivors. Few prognostic tests are available to predict PTB. A short transvaginal ultrasound cervical length (TVU CL) has been shown to be a good predictor of PTB.

Other strategies have been adopted for prevention of PTB. The evidence supports the use of vaginal progesterone in singleton pregnancies with short cervix.

However, the predictive value of the research has recently been questioned, as the threat rate from preterms in the low-risk population has not decreased over time. Numerous clinical studies have been conducted to improve and identify effective prevention strategies in the threat of preterm birth. Among the parameters studied, in addition to the measurement of the uterine cervix and its complaints during the three trimesters of pregnancy, an evaluation of the cervical consistency index (CCI) was also proposed, i.e. an ultrasound evaluation of cervical softness.

DETAILED DESCRIPTION:
Numerous clinical studies have been conducted to improve and identify effective prevention strategies in the threat of preterm birth. Among the parameters studied, in addition to the measurement of the uterine cervix and its changes during the three trimesters of pregnancy, the evaluation of the cervical consistency index (CCI), or an ultrasound evaluation of cervical softness, was also proposed.

Reduced CCI values correspond to greater compressibility and cervical softness. Studies conducted to study cervical remodeling on animal models suggest an early increase in cervical softness that begins immediately after conception followed by shortening and dilation in the terminal stages of pregnancy so that minimal changes in cervicometry correspond to a significant increase in cervical softness . Therefore the study of the early stages of cervical remodeling, such as cervical softness through the ICC, could allow to identify in a timely manner women with an increased risk of preterm birth.

The purpose of this study is to define and standardize the transvaginal technique to determine the CCI, its reference range and establish its potential predictive use in the threat of preterm birth before 32, 34 and 37 weeks.

The purpose of this study is to verify the hypothesis that the introduction of a universal screening program with TVU CL and CCI measurement, in the three trimesters of pregnancy, may be associated with a predictive ability to deliver preterm higher than current protocols.

ELIGIBILITY:
Inclusion Criteria:

Singleton gestations 18-50 years of age

Exclusion Criteria:

Multiple gestation Ruptured membranes or fetal structural or chromosomal abnormality at the time of randomization Labor or cerclage in situ at the time of randomization Women with altered state of consciousness, seriously ill, with mental handicaps;

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 500 (Estimated)
Dates: Start 2020-04-25 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Preterm delivery | Less than 37 weeks gestation

SECONDARY OUTCOMES:
Gestational age at delivery | Time of delivery
Preterm birth rates | Less than 24, 28, 34 weeks gestation
Birth weight | Time of delivery
Low birth weight | Time of delivery
  Birth weight <2500g
Neonatal death | Between birth and 28 days of age
Composite adverse neonatal outcome | Between birth and 28 days of age
  Includes necrotizing enterocolitis, intraventricular hemorrhage (grade 3 or higher), respiratory distress syndrome, bronchopulmonary dysplasia (BPD), retinopathy, blood-culture proven sepsis and neonatal death
Admission to neonatal intensive care unit | Between birth and 28 days of age

CONTACTS AND LOCATIONS:
Overall Officials: Fabiana Savoia, MD, Principal Investigator — University of Campania Luigi Vanvitelli; Maddalena Morlando, MD, Study Chair — University of Campania Luigi Vanvitelli
Locations (1):
- University of Campania "Luigi Vanvitelli", Naples, Italy

IPD SHARING:
Plan to Share IPD: No